CLINICAL TRIAL: NCT05435417
Title: Effect of Segmentation Techniques (Manual Versus Semiautomatic) on the Accuracy of the Reconstructed Mandibular Condyle Using CBCT(A Diagnostic Accuracy Study)
Brief Title: Effect of Segmentation Techniques (Manual Versus Semiautomatic) on the Accuracy of the Reconstructed Mandibular Condyle Using CBCT
Acronym: CBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas El Saket, principle investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RAD 7:1-1
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Segmentation Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual segmentation technique of CBCT images of the condyles. (Experimental): Using the manual edition built in tool, first a brush of small size will be used to demarcate the outline of the condyle in the sagittal cuts. Then shading the demarcated condylar area with a brush of larger size in each slice. The outline of the condyle will be refined on all cuts. The software built in tool 'create surface' will be used to create the segmented 3D volume
  Interventions: Radiation: CBCT radiation
- Semiautomatic segmentation technique of CBCT images of the condyles. (Experimental): Using the water shed built in tool, first a brush of small size will be used to demarcate the outline of the condyle by the 'background' option in all planes. Then using the 'foreground' option, a brush of larger size will be used to shade the condylar area. The software built in tool 'expand water shed' will be used to include the whole condyle. At last, 'create surface' option will be used to create the segmented 3D volume.
  Interventions: Radiation: CBCT radiation
- Actual physical measurements of the condyles on the dry mandibles (No Intervention): For linear measurements, actual physical measurements will be done on the dry mandibular condyles, using digital caliper, as mentioned before.
  For volumetric measurements, water displacement technique will be used. The mandibular condyle will be immersed in a graduated beaker containing water till the level of the glued gutta percha. The volume of the displaced water will be measured and will represent the actual volume of the condyle

INTERVENTIONS:
Radiation: CBCT radiation — CBCT scanning
  Arms: Manual segmentation technique of CBCT images of the condyles.; Semiautomatic segmentation technique of CBCT images of the condyles.

SUMMARY:
Effect of Segmentation Techniques (Manual versus Semiautomatic) on the Accuracy of the Reconstructed Mandibular Condyle using CBCT

DETAILED DESCRIPTION:
It will be used to segment the mandibular condyle and asses its volumetric and linear measurements. Therefore, the accuracy of the segmentation techniques of the mandibular condyle will be determined

ELIGIBILITY:
Inclusion Criteria:

* Intact dry human skulls and mandibles.

Exclusion Criteria:

* Presence of fracture, pathological lesions, or skeletal deformities in the condylar area.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Linear assessment of the condyles | one month
  Linear measurements will be calculated in millimeters by Built-in measuring tool (ruler) in the software + digital caliper on the dry mandibles

SECONDARY OUTCOMES:
Volumetric assessment of the condyles | one month
  For volumetric measurements, the volume of the segmented condyle, either by manual or semiautomatic segmentation technique, will be automatically calculated by the software. Volumetric measurements will be calculated in cubic millimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt